CLINICAL TRIAL: NCT04891341
Title: Investigation of the Effects of Technology Supported Different Physiotherapy Approaches on Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Mert Doğan, Physiotherapist in Neurological Rehabilitation Department, Master of Science, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-53875521-050-713
Record Dates: First submitted 2021-05-02; First posted 2021-05-18 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Multiple Sclerosis
Keywords: Virtual Reality; Telerehabilitation; Task-oriented Circuit Therapy; Kinematics; Kinematic Analysis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology Supported Task-Oriented Circuit Therapy Group (Experimental): Ten workstations, which are frequently used in the literature and determined according to the clinical experience of the research team, have been created. Each workstation will be applied for a total of 1 hour, in the form of 5 minutes of training and 1 minute of rest.
  Interventions: Other: Technology Supported Task-Oriented Circuit Training
- Home-based Telerehabilitation Group (Active Comparator): To the telerehabilitation group; A home program consisting of strengthening, balance and coordination exercises determined according to the needs of volunteers with MS will be given. A session will be applied in the home program under the guidance of a physiotherapist. The exercise will take 1 hour. The exercise participation status of the patient will be monitored with a mobile (smartphone) application. Exercises will be constantly updated according to the needs of the patient, the updated exercises will be sent to the mobile application via video, and the patient will be able to communicate with the physiotherapist via video conference whenever he / she wishes. Progress and complication of the treatment program will be achieved by increasing the weights used, changing the ground characteristics and support surface during balance exercises and increasing the complexity of coordination exercises.
  Interventions: Other: Home-based Telerehabilitation

INTERVENTIONS:
Other: Technology Supported Task-Oriented Circuit Training — Ten workstations, which are frequently used in the literature and determined according to the clinical experience of the research team, have been created. Each workstation will be applied for a total of 1 hour, in the form of 5 minutes of training and 1 minute of rest.
  1. Sit to stand
  2. Standing and trunk training
  3. Standing and lower limb training
  4. Stepping
  5. Walking
  6. Walking with object manipulation
  7. Climbing and descending stairs
  8. Unilateral upper extremity activity training (VR)
  9. Bilateral upper extremity activity training (VR)
  10. Upper extremity reaction time training (VR) Virtual reality games will be played using the USE-IT intelligent physiotherapy game system. The system offers unilateral, bilateral and bimanual upper extremity training to individuals with a 55 inch touch screen and 7 computer games (balloon popping, car washing, plumbing, arithmetic, apartment, drum and matching).
  Arms: Technology Supported Task-Oriented Circuit Therapy Group
Other: Home-based Telerehabilitation — Strengthening, balance and coordination exercises will be sent to the participants via a mobile application. Patients will do the exercises at home and send a notification to their physiotherapist. Intervention will be applied for 1 hour, 3 days a week for 8 weeks.
  Arms: Home-based Telerehabilitation Group

SUMMARY:
Multiple Sclerosis (MS) is an autoimmune disease characterized by chronic inflammation, demyelination and axonal loss of the central nervous system. The etiology of the disease is not known exactly and possible causes are; genetic, vitamin D deficiency, viral, environmental and autoimmune factors have been identified. Common findings of MS are in the literature; sensory, visual problems, fatigue, urinary retention / incontinence, motor problems (inability to walk, upper extremity skills, coordination and balance problems), cognitive deficits, tone, speech and swallowing disorders. In the rehabilitation of MS; It is seen that balance, coordination, strengthening, aerobic and neurodevelopmental exercise methods are used and these approaches have reached moderate / high level evidence in the literature. Task-oriented circuit therapy(TOECT), one of the current neurophysiology-based approaches; It is a motor learning-based exercise approach based on the theory of dynamic systems, one of the theories of motion control, aiming at the acquisition of skills for a specific functional activity. When the existing studies are examined, it has been determined that there are a limited number of randomized controlled studies examining the effects of TOECT and that sufficient evidence cannot be obtained with these studies. In previous studies, it has been observed that standardization of exercise approaches applied to the control group could not be achieved and the control groups generally included applications that could create passive or effect summation compared to the experimental groups. In addition, in the literature, TOECT, which includes rehabilitation games to be applied in the form of station training, in MS patients; There is no randomized controlled study examining the effects on balance, walking, fatigue, trunk and upper extremity functions and kinematics. In this direction, the purpose of the research is; To examine the effects of technology-supported TOECT and technology-supported home program applied as station training on walking, quality of life, fatigue, balance, trunk and upper extremity functions of patients with MS, using kinematic and clinical methods. Volunteers who agree to participate in the study will be divided into two groups by the block randomization method. Both groups will receive exercise training 3 sessions per week (24 sessions in total) for 8 weeks. Evaluations will be made before and after 8 weeks treatment

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Relapsing Remitting, Primary Progressive or Secondary Progressive MS according to McDonald criteria,
* Between the age of 18 and 50 years
* EDSS score greater than 2, less than 5.5,
* Mini Mental State Test score of 24 and above,
* Volunteers who have access to smartphone (mobile phone) through themselves or their relatives will be included in the study.

Exclusion Criteria:

* Surgery or botox application for spasticity in the last 6 months,
* Having an attack history in the last 3 months,
* Received physical therapy and rehabilitation services in the last 6 months,
* Any pain in any part of the body, previous surgery, any orthopedic problem,
* Have a secondary neurological, orthopedic or systematic condition that prevents standing independently,
* With severe peripheral vestibular involvement,
* EDSS- Pyramidal functions score equal to and greater than 4,
* Patients who do not agree to participate in the study and do not give written consent will not be included in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-07-16 (Actual); Study Completion 2022-07-17 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | Change between baseline and after 8 weeks treatment.
  Berg Balance Scale will be used to determine the balance exposure level of the volunteers. It is a scale that includes the performance of 14 different tasks between 0 (not applicable) and 4 (normal performance). In this scale, which is evaluated over 56 points; Scores between 0 and 20 indicate imbalance, scores between 21 and 40 indicate that the balance is acceptable, and scores between 41 and 56 indicate that the balance is good.
Multiple Sclerosis Quality of Life Scale (MSSQL-54) | Change between baseline and after 8 weeks treatment
  Individuals' quality of life will be evaluated with MSQOL-54. In this scale consisting of 12 chapters and 54 questions in total, physical function, social function, physical role limitations, emotional role limitations, cognitive function, pain, emotional state, energy, sexual function, health perception, general quality of life, health stress and emotional well-being.

SECONDARY OUTCOMES:
Trunk Impairment Scale | Change between baseline and after 8 weeks treatment.
  Trunk Impairment Scale will be used to evaluate the volunteers' trunk control. The scale consists of 17 items, 3 of which are related to static balance, 10 to dynamic balance, and 4 to the coordination ability of the stabilizer muscles. The scale is in the range of 0-23 points. High scores indicate good trunk control.
Timed Up and Go Test | Change between baseline and after 8 weeks treatment.
  The Timed Get Up and Go Test will be used to evaluate the volunteers' functional mobility skills. Volunteers are asked to sit on a chair. A cone is placed 3 meters away from the chair in a linear fashion. The volunteer is asked to get up, walk around the cone and sit back on the chair. The time to complete this task will be recorded by measuring with a stopwatch. The test will be repeated 3 times and the average time will be noted.
Goal Assesment Scale | Change between baseline and after 8 weeks treatment.
  This scale, which is widely used in patient-centered treatment approaches, includes the creation of the goal that the patient wants to reach as a result of the treatment, by the physiotherapist and the patient. The expected result is initially set as "0", -2 means the worst expected result, while +2 represents the most positive possible result.
  Fatigue Intensity Scale: Fatigue intensity scale will be used to evaluate fatigue. The scale consists of 9 items. Each item is rated from 1 to 7. The score of the scale is obtained by the arithmetic mean of all items. People with a score of 4 and above are considered to be tired.
ABILHAND-Stroke | Change between baseline and after 8 weeks treatment.
  ABILHAND Stroke Hand Function Questionnaire will be used to question the hand functions of volunteers. In the questionnaire, the level of difficulty perceived by the volunteers while performing activities such as feeding, dressing and housework is questioned. The questionnaire consists of 56 items and each item is scored as 0 (impossible), 1 (difficult) and 2 (easy). High score means good hand skills.
Minnesota Manual Dexterity Test | Change between baseline and after 8 weeks treatment.
  Minnesota Manual Dexterity test will be used to evaluate volunteers' hand agility. Test 60 blocks; There are two stages of placement and translation. The placement test is performed by the volunteer placing the blocks towards the distance from the target close to him, and the total time is recorded. The placement test will be repeated for both hands. In the flip test, the volunteer is asked to take the blocks from the corner of the dominant side with the non-dominant hand, turn them bimanually and place them with the dominant side. The test goes from the far dominant corner to the non-dominant corner. The second row starts on the non-dominant side and runs towards the dominant side. At this stage, the person takes the block with the dominant hand, turns it bimanually and places it with the non-dominant side. This is repeated in the third and fourth rows as in the first and second rows and the total time is recorded. In the literature, it is recommended for use in patients with MS.
Twelve Item MS Walking Scale | Change between baseline and after 8 weeks treatment.
  This 12-item scale evaluates the limitations of the MS patient in walking in the last two weeks. Scoring is made between 1-5. In this questionnaire, in which the patient evaluates his own walking performance, a high score indicates that walking ability is affected or the patient has difficulty in walking.
Kinematic Analysis During Functional Activities | Change between baseline and after 8 weeks treatment.
  XSENS MVN-Awinda sensors will be used to measure volunteers' joint angles in different functions. This sensor system is frequently used in the literature for motion analysis. Joint angles will be measured using sensors during the following activities:
  1. Walking
  2. Functional reaching,
  3. Sit to Stand
  4. Touch the middle of the head,
  5. Hanging jackets,
  6. Eating,
  7. Touch the back pocket of your trousers,
  8. Get the phone to ear. Tests other than walking and standing up without sitting will be performed bilaterally. The materials used during the tests will be in the same physical properties and conditions for all patients.
International Cooperative Ataxia Rating Scale | Change between baseline and after 8 weeks treatment.
  The scale consists of 4 sub-parameter: posture and gait disturbances, kinetic functions, speech and oculomotor disorders. Posture and gait disturbances sub-parameter consists of 7 questions 34 points, kinetic functions 7 questions 52 points, speech disorders 2 questions 8 points, oculomotor disorders 3 questions 6 points. The score range is 0-100, and higher scores indicate increased disease severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Mert Doğan, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided